CLINICAL TRIAL: NCT02102282
Title: Observational Study of Breast Cancer Diagnosed During Pregnancy
Brief Title: Breast Cancer During Pregnancy
Acronym: BRCAPRE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PR(AMI)83/2012
Record Dates: First submitted 2014-03-29; First posted 2014-04-02 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-03

CONDITIONS: Pregnancy; Breast Cancer
Keywords: Pregnancy; Breast Cancer; Chemotherapy; Surgery; Obstetric managment
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and tissue samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subject study: Patients with breast cancer during pregnancy

SUMMARY:
Patients are managed clinically according to ad hoc standards and scientific knowledge by a multidisciplinary team. Clinical decisions are made after a patient physician discussion. Blood and tissue samples are collected. Diagnostic, obstetric management surgical treatment, systemic treatment, perinatal results and follow up data are collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients with breast cancer diagnosed during pregnancy

Exclusion Criteria:

* Patients who refuse informed consent

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with breast cancer diagnosed during pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2012-10; Primary Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Perinatal results | Delivery
  Gestational age, weight, Apgar, blood tests

SECONDARY OUTCOMES:
Maternal outcome | 5 year and 10 year
  Over all survival, disease free survival

CONTACTS AND LOCATIONS:
Overall Officials: Octavi Cordoba, PhD MD, Principal Investigator — Hospital Vall d'Hebron
Locations (1):
- Hospital Vall d'Hebron, Barcelona, Spain

REFERENCES:
- [Result] Cordoba O, Llurba E, Saura C, Rubio I, Ferrer Q, Cortes J, Xercavins J. Multidisciplinary approach to breast cancer diagnosed during pregnancy: maternal and neonatal outcomes. Breast. 2013 Aug;22(4):515-9. doi: 10.1016/j.breast.2012.10.005. Epub 2012 Oct 30. PMID 23116970
- [Result] Cordoba O, Llurba E, Cortes J, Sabadell MD, Lirola JL, Ferrer Q, Xercavins J. Complete pathological remission in a patient with hormone-receptor positive and c-erbB-2 expression-negative breast cancer treated with FAC chemotherapy during pregnancy. Tumori. 2010 Jul-Aug;96(4):629-32. doi: 10.1177/030089161009600420. PMID 20968147